CLINICAL TRIAL: NCT04109846
Title: Transfer of Aneuploid or Mosaic Embryos Following Preimplantation Genetic Testing
Brief Title: Pregnancy and Developmental Outcomes After Transfer of Reportedly Aneuploid or Mosaic Embryos
Acronym: TAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ruth Bunker Lathi, Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-46420
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Aneuploidy; Mosaicism; Pregnancy Outcome
Keywords: Preimplantation Genetic Testing for Aneuploidy; Preimplantation Genetic Screening; embryo transfer; mosaic; aneuploid
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Intervention Model Description: Patients desiring frozen embryo transfer or aneuploid or mosaic embryo. Patients will be counseled regarding risks and obstetric and pediatric outcomes will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-euploid Transfer (Experimental): Patients desiring pregnancy who have no acceptable euploid embryos available for transfer who chose to undergo embryo transfer of a non-euploid embryo (either aneuploid or mosaic).
  Interventions: Other: Non-euploid embryo transfer
- Euploid Transfer (Active Comparator): Patients desiring pregnancy who are undergoing euploid embryo transfer
  Interventions: Other: Euploid Transfer

INTERVENTIONS:
Other: Non-euploid embryo transfer — Other than choice of embryo for transfer, all other medical interventions will be standard of care protocols
  Arms: Non-euploid Transfer
Other: Euploid Transfer — Standard of Care Protocol
  Arms: Euploid Transfer

SUMMARY:
To determine how often embryos reported to be abnormal by preimplantation genetic testing result in liveborn infants. To evaluate whether the pregnancies that result from these embryos are higher risk for complications and whether the resulting babies have higher risk for health or developmental issues in the first five years after birth.

DETAILED DESCRIPTION:
Genetic testing modality and results will be recorded

Pregnancy per transfer will be recorded

Patients in the study agree to provide medical records of their pregnancy.

Any genetic testing or fetal testing will be carefully reviewed and recorded by the study team.

For patients with live births, pediatric records will be collected for up to 5 years.

As well as surveys for developmental milestones.

There is no financial compensation for study participants

ELIGIBILITY:
Inclusion Criteria:

* Available aneuploid or mosaic embryos
* No other acceptable embryos available
* Willing to travel to Stanford for treatment
* English language fluency

Exclusion Criteria:

* Use of international donor eggs or sperm not tested according to FDA guidelines.
* Living outside the United States
* Embryos with Triploidy are not eligible for transfer in this protocol

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2035-04 (Estimated); Study Completion 2039-04-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Rate | 3 years
  Number participants who undergo embryo transfers that lead to a positive pregnancy test

SECONDARY OUTCOMES:
Live birth rate | 4 years
  Number participants who conceive after embryo transfer and have a live birth.
Obstetric complications | 4 years
  Number of participants who have a maternal of fetal complication after embryo transfer
Pediatric Development | 7 years 3 months
  Number of newborns and children who have abnormal pediatric development at 3 months, 2 years and 5 years following birth

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Lathi, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Fertility and Reproductive Medicine Center, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will only reported in aggregate

REFERENCES:
- [Background] Munne S, Spinella F, Grifo J, Zhang J, Beltran MP, Fragouli E, Fiorentino F. Clinical outcomes after the transfer of blastocysts characterized as mosaic by high resolution Next Generation Sequencing- further insights. Eur J Med Genet. 2020 Feb;63(2):103741. doi: 10.1016/j.ejmg.2019.103741. Epub 2019 Aug 21. PMID 31445143
- [Background] Victor AR, Tyndall JC, Brake AJ, Lepkowsky LT, Murphy AE, Griffin DK, McCoy RC, Barnes FL, Zouves CG, Viotti M. One hundred mosaic embryos transferred prospectively in a single clinic: exploring when and why they result in healthy pregnancies. Fertil Steril. 2019 Feb;111(2):280-293. doi: 10.1016/j.fertnstert.2018.10.019. PMID 30691630
- [Background] Zhang L, Wei D, Zhu Y, Gao Y, Yan J, Chen ZJ. Rates of live birth after mosaic embryo transfer compared with euploid embryo transfer. J Assist Reprod Genet. 2019 Jan;36(1):165-172. doi: 10.1007/s10815-018-1322-2. Epub 2018 Sep 24. PMID 30246223
- [Background] Munne S, Blazek J, Large M, Martinez-Ortiz PA, Nisson H, Liu E, Tarozzi N, Borini A, Becker A, Zhang J, Maxwell S, Grifo J, Babariya D, Wells D, Fragouli E. Detailed investigation into the cytogenetic constitution and pregnancy outcome of replacing mosaic blastocysts detected with the use of high-resolution next-generation sequencing. Fertil Steril. 2017 Jul;108(1):62-71.e8. doi: 10.1016/j.fertnstert.2017.05.002. Epub 2017 Jun 1. PMID 28579407
- [Background] Greco E, Minasi MG, Fiorentino F. Healthy Babies after Intrauterine Transfer of Mosaic Aneuploid Blastocysts. N Engl J Med. 2015 Nov 19;373(21):2089-90. doi: 10.1056/NEJMc1500421. No abstract available. PMID 26581010
- See also: Stanford Fertility Research website — https://www.stanfordchildrens.org/en/services/fertility-and-reproductive-health/clinical-trials-and-research/tame.html